CLINICAL TRIAL: NCT07118241
Title: A PHASE II PROSPECTIVE RANDOMIZED DOUBLE-MASKED CONTROLLED STUDY ASSESSING THE SAFETY & EFFICACY OF RHPRG4 (450 µG/ML RECOMBINANT HUMAN PROTEOGLYCAN 4) COMPARED TO VEHICLE FOR THE TREATMENT OF SJÖGREN'S RELATED DRY EYE DISEASE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lubris Bio Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHPRG4-SJÖGREN'S-002
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sjögren's Syndrome
Keywords: Sjogrens Syndrome; Dry Eye
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vehicle Control (Placebo Comparator): PBS Based Vehicle Control
  Interventions: Drug: Vehicle Control
- rhPRG4 450ug/ml (Experimental): rhPRG4 450ug/ml
  Interventions: Drug: Recombinant Human Proteoglycan 4

INTERVENTIONS:
Drug: Recombinant Human Proteoglycan 4 — rhPRG4 450ug/ml
  Arms: rhPRG4 450ug/ml
Drug: Vehicle Control — PBS based Vehicle Conrtol
  Arms: Vehicle Control

SUMMARY:
rhPRG4-Sjögren's-002 is a prospective multi-center study conducted in Australia to evaluate the safety and efficacy of topically-applied rhPRG4 in subjects with Sjögren's related Dry Eye Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to comprehend and provide a signed and dated consent form.
2. Are 18-75 years at time of consent;
3. Have been diagnosed with SS for at least 3 months prior to ICF;
4. Have been using artificial tears as the only topical treatment of SS related dry eye for at least 30 days prior to Visit 1;
5. Have been stably using systemic medications for at least one month prior to Visit 1;
6. Have Global SANDE score ≥ 40;
7. Average VAS score for typical symptoms of dry eye (dryness, foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia) ≥ 25 mm, none < 5 mm;
8. Have Oxford corneal fluorescein staining grade of ≥ 1 and ≤ 2 in each eye (OD & OS both ≥ 1 and ≤ 2);
9. Stated willingness to comply with all study procedures, attend all scheduled clinic visits, and continue participation for the duration of the study.
10. Ability to self-administer study medication and willingness to adhere to the medication regimen.

Exclusion Criteria

1. Are currently or have a history of any ocular or systemic disorder or condition other than dry eye that based on investigator judgment will interfere with the interpretation of the study results. Examples of ocular or systemic disorders or conditions include active ocular infection, conjunctivochalasis, superior limbic keratoconjunctivitis, limbal stem cell deficiency, allergic conjunctivitis, giant papillary conjunctivitis, atopic keratoconjunctivitis, anterior basement membrane dystrophies, neurotrophic keratitis, corneal dystrophy, exposure keratitis, moderate to severe blepharitis, ocular trauma, progressive or degenerative corneal conditions, uveitis, and systemic infection;
2. Have used any topical ocular medications (other than artificial tears), therapeutic medical devices, or undergone ocular surgery within the 30 days prior to Visit 1. Topical ocular medications include cyclosporine, lifitegrast, corticosteroid eye drops, and autologous/serum. Therapeutic medical devices include trigeminal stimulation, meibomian glad warming (excepting at home masks) or expression, intense pulsed light, low level light therapy, etc. Ocular surgeries include laser or refractive surgical procedures, insertion of punctal or punctal cauterization;
3. Are unwilling to forgo the use of topical medications (other than IMP and limited artificial tear use), medical devices or ocular surgery from Visit 1 through Visit 4.
4. Have only one eye;
5. Are unwilling to adhere to t.i.d. administration of vehicle during run-in;
6. Are unwilling to limit the use of artificial tears to no more than 4 days during run-in;
7. Have begun regularly using systemic compounds for SS or SS-related dry eye during the one month prior to Visit 1. Systemic compounds include omega-3 oil (fish oil, flaxseed oil, etc.), systemic corticosteroids, immunosuppressants, and biologics that based on investigator judgment will interfere with the interpretation of the study results.
8. Are unwilling to maintain a stable regimen of systemic compound use during the duration of the study;
9. Have known hypersensitivity to one of the components of the study or procedural medications;
10. Have participated in another clinical study at the same time as the present study or within 30 days of Visit 1;
11. Have a history of drug, medication or alcohol abuse or addiction;
12. Are females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) who meet any one of the following conditions:

    1. are currently pregnant or,
    2. have a positive result on the urine pregnancy test at the Screening Visit or,
    3. intend to become pregnant during the entire course of and 30 days after the study treatment periods, or,
    4. are breast-feeding or,
    5. not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods, during the entire course of and 30 days after the study treatment periods;
13. Are males with a female partner of child bearing potential where:

    1. the male is not surgically sterilized or,
    2. where the male partner cannot provide information regarding the female partner's child bearing status or,
    3. where the child bearing status of the female partner does not meet that of Exclusion Criteria 12; however, the female partner of a male participant will not be required meet Exclusion Criteria 12b.
14. Have a history of a serious physical or psychiatric disorder that, in the investigator's opinion, could prevent compliance with study procedures or affect study participation;
15. Have any other surgical or medical condition or finding that in the opinion of the investigator would compromise the subject's safety or participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of rhPRG4 by looking at the frequency of patients attaining complete resolution of total corneal staining with fluorescein (Oxford Scale) at Day 28 | From baseline to the end of treatment at day 28
  To assess the efficacy of rhPRG4 by looking at the frequency of patients attaining complete resolution of total corneal staining with fluorescein (Oxford Scale) at Day 28

SECONDARY OUTCOMES:
To assess the safety of rhPRG4 by observation of the severity of treatment-emergent adverse events for the study duration | From baseline to day 28
  To assess the safety of rhPRG4 by observation of the severity of treatment-emergent adverse events for the study duration
To assess the safety of rhPRG4 by observation of the change in BCVA over 28 days | From baseline to day 28
  To assess the safety of rhPRG4 by observation of the change in BCVA over 28 days
To assess the safety of rhPRG4 by observation of signs evaluated by slit lamp examination (SLE) (Meibomian glands, Eyelid Erythema, Eyelid Oedema, Lashes, Conjunctiva Erythema, Lens, Iris, Anterior Chamber, Hyperemia, Corneal transparency & Corneal neo | From baseline to day 28
  To assess the safety of rhPRG4 by observation of signs evaluated by slit lamp examination (SLE) (Meibomian glands, Eyelid Erythema, Eyelid Oedema, Lashes, Conjunctiva Erythema, Lens, Iris, Anterior Chamber, Hyperemia, Corneal transparency & Corneal neovascularization)
To assess the safety of rhPRG4 by observation of intraocular pressure (IOP) | From baseline to day 28
  To assess the safety of rhPRG4 by observation of intraocular pressure (IOP)
To assess the efficacy of rhPRG4 using the total VAS score for dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia (anchors: none & severe) at Day 28 | From baseline to day 28
  To assess the efficacy of rhPRG4 using the total VAS score for dryness, foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision and photophobia (anchors: none & severe) at Day 28
To assess the efficacy of rhPRG4 using the SANDE score compared to vehicle at Day 28 | From baseline to day 28
  To assess the efficacy of rhPRG4 using the SANDE score compared to vehicle at Day 28
To assess the efficacy of rhPRG4 using the Oxford staining score, both per eye and as a total score per subject compared to vehicle at Day 28 | From baseline to day 28
  To assess the efficacy of rhPRG4 using the Oxford staining score, both per eye and as a total score per subject compared to vehicle at Day 28

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Univ of New South Wales, Sydney, New South Wales
  - OTA, Brisbane, Queensland
  - Queensland University of Technology, Brisbane, Queensland
  - University of the Sunshine Coast, Maroochydore, Queensland
  - University of Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided